CLINICAL TRIAL: NCT02065596
Title: Hematopoietic Stem Cell Transplant for Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE12Z13
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia; SCD
Keywords: Sickle Cell Disease; Sickle Cell Anemia; GvHD; fludarabine
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — fludarabine; fludarabine phosphate; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Immunomodulation with Fludarabine prior to HSCT (Experimental): Fludarabine given beginning at 25mgm/m2 three times per day. Patients may be escalated up to 25mgm/m2 five times per day depending on dose-limiting toxicity
  Interventions: Drug: Fludarabine; Procedure: Hematopoietic Stem Cell Transplant (HSCT)

INTERVENTIONS:
Drug: Fludarabine — the study will begin with enrollment of an initial safety cohort of at least 10 subjects at the lowest dose, after which enrollment will pause until the dose-limiting toxicity (DLT) period has been completed. If a patient experiences DLT, defined as failure to engraft. In which case, the patient may be advanced to two higher doses.
  Other Names: Fludarabine monophosphate
Procedure: Hematopoietic Stem Cell Transplant (HSCT) — Three weeks after Immunomodulation patients will be infused with matched bone marrow from a sibling, unrelated donor, haploidentical donor, or cord blood. Patients will be followed for the following year.

SUMMARY:
This is a study of patients with sickle cell disease. It aims to find out if people with sickle cell disease can be cured by changing their immune system before they have blood stem cell transplants. Doctors will give patients a new drug (fludarabine) to see if this drug changes patients immune system and reduces the patient's cells (host) from rejecting donor cells (graft) after the patient gets a Hematopoietic (blood) stem cell transplant.

DETAILED DESCRIPTION:
Primary Objective

1. To evaluate the safety and feasibility of hematopoietic stem cell transplant (HSCT) after treatment with fludarabine in adult patients with Sickle Cell Disease (SCD).

Secondary Objective(s), in HSCT for SCD

1. To evaluate the rates of disease-free and overall survival in both MSD and alternate graft donor (MUD, haploidentical, or cord blood-derived) recipients
2. To evaluate fertility in matched sibling and alternate-donor graft recipients
3. To evaluate GVHD rates in MSD and Alternate Graft Donor recipients in SCD.
4. To evaluate cerebral, pulmonary, renal, and generalized vasculopathy before and after HSCT in SCD.
5. To evaluate hematopoiesis and erythropoiesis before and before HSCT in SCD.
6. Modulation of SCD Phenotype by Allogeneic Transplantation. Rigorous clinical follow-up will be performed, per routine care, to evaluate those consequences of SCD that will be modified by allogeneic transplantation in the short-term (4-12 weeks), in the medium-term (12-24 weeks) and in the long-term (>24 weeks). Short-term changes would include disappearance of stress hematopoiesis and erythropoiesis; medium- and long-term changes would include effects on pain, fertility (TSH, LH), cognition (routine cognitive assessments), and end-organ damage (including urine albumin-to-creatinine ratios and tricuspid regurgitant jet velocities, as indicated).

Procedures:

The study will start with at least 10 and up to 25 patients. They will be given the lowest starting dose of fludarabine. This is done to make sure it is safe. Researchers will watch the patients during what is called the dose-limiting toxicity (DLT) period. Their safety will be monitored by a Safety Monitoring Committee, which is made up of people who run research studies. The study will not take new patients until the DLT period is done.

If at least 3 of the 10 patients enrolled do not benefit, the maximum tolerated dose (MTD) will be considered exceeded. After the DLT period is complete, patients will receive a stem cell transplant from a genetically matched donor. Patients will be continued to be monitored for a year after the transplant.

To prepare for the transplant patients will have to undergo the following treatments:

* an exchange transfusion
* a stem cell graft infusion from either a:

  * perfectly matched sibling donor (called MSD),
  * perfectly matched but unrelated donor (called MUD),
  * a half-matched related donor (called Haploidentical), or
  * a cord blood donor
* rabbit antithymocyte globulin (ATG)
* cytoxan (a type of chemotherapy)
* Fludarabine (you get this medicine a few weeks before transplant and again, as part of the routine chemotherapy treatment). This is the main drug being studies in this research
* total body irradiation (also called TBI)
* tacrolimus, mycophenolate (MMF) and/or methotrexate (MTX). These drugs will weaken your immune system. They are given to lower your chances of getting GVHD and rejecting the donor cells.

Patients will be in the study for approximately 14 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following inherited hemoglobin gene disorders:

  * a. Hemoglobin SS
  * b. Hemoglobin SC
  * c. Hemoglobin S-Beta-zero-Thalassemia or
  * d. Hemoglobin S-Beta-plus Thalassemia with an episode of multi-organ failure within 5 years of eligibility

Patients must meet one of the following risk criteria:

* Low Risk (Red Light. Stop and consider therapy closely): Must have matched sibling donor grafts, failed conventional therapy as determined by the PI, and evidence for morbid disease (one of the following):

  * a. 2 or more painful episode/year (requiring Emergency Department or inpatient care) x 2 years or
  * b. 1 or more diagnoses of Acute Chest Syndrome within 5 years, or
  * c. 2-year mortality 5-10% or
  * d. Baseline LDH>600 IU or
  * e. History of sepsis, with or without a WBC>13.5, or
  * f. On chronic transfusions
* Moderate Risk (Yellow Light. Reasonable to proceed, but with caution): May have alternate donor grafts (haploidentical or matched unrelated donor), if MSD is not available. Must have history of high-level vasculopathy, as defined by at least one of the criteria below:

  * a. Urine Albumin to Creatinine Ratio of >300mg/g or eGFR 50-90 ml/min x 2 evaluations within 3 months or
  * b. History of overt clinical stroke, or progressive cerebral vasculopathy radiographically or
  * c. 1 or more diagnoses of Acute Chest Syndrome, multi-organ failure, or sickle hepatopathy within 7 years, or
  * d. Excessively morbid disease manifest as VOCs at a rate of 2 or more per year x 2-years or uncontolled retinal disease attributed to SCD. These patients can be considered for moderate-risk alternate donor transplants. The palliative nature of the transplant will be explicit in the consent.
  * e. 2-year mortality >10-15%

    * i. Baseline WBC>13.5 and on chronic transfusions or baseline LDH>600 or age >35 years old,
    * ii. Baseline TRV ≥3 m/s,
    * iii. Chronic transfusion therapy and age >35 years old or male gender,
    * iv. Baseline LDH>600 and age >35 years old or history of sepsis
    * v. History of sepsis and age >35 years old or male gender.
  * f. History of multi-organ failure
* High Risk (Green light, proceed if possible): All donor types are eligible. Must have high risk disease and a >15% risk of 2-year mortality as defined by at least one of the criteria below.

  * a. Baseline TRV ≥3 m/s and baseline WBC >13.5 or on chronic transfusions or history of sepsis or age >35 years old,
  * b. Baseline WBC>13.5 and chronic transfusions or baseline LDH>600 or age >35 years old
  * c. Age >35 years old and chronic transfusions

To determine eligibility as a bone marrow transplant patient:

* Available suitable donor

  * a. 6/6 HLA-matched sibling donor (HLA A, B, and DRB1), bone marrow only
  * b. 8/8 HLA-matched unrelated donor (HLA A, B, C, DRB1), bone marrow only
  * c. 4/8, 5/8, 6/8, 7/8 Haploidentical donor, bone marrow only
* Patients must have adequate hematologic, hepatic, and renal function as defined below:

  * Direct bilirubin within 3 X normal institutional limits
  * ALT (SGPT) < 3 X institutional upper limit of normal
  * Creatinine clearance >21 mL/min/1.73 m^2 for subjects with creatinine clearance values below 50 mL/min/1.73 m^2, the principal investigator may use discretion for appropriate fludarabine dose adjustment as noted.
  * Patients must have adequate pulmonary function as defined by Pulmonary function: DLCO r40% (adjusted for hemoglobin) and FEV1r50%.
* Contraception/Child Bearing The effects of Fludarabine, cytoxan, ATG, tacrolimus/sirolimus and MTX are cumulatively known to be deleterious to the health of the developing human fetus. For this reason, and because of teratogenic potential, all women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) for the duration of study participation and for 12 months after completing treatment.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Red cell alloimmunization to a degree that precludes extended transfusion
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Subjects must not have evidence of impaired liver function due to iron overload, +/- hepatitis. Patients will be evaluated by liver consult if ferritin >1500, history of hepatitis,or ALTis ≥3 X Upper limit of normal (ULN). Recommended evaluations could include liver biopsy if there is evidence for significant hepatic iron deposition or fibrosis/cirrhosis on T2* MRI of the liver.
* eGFR <21 ml/min
* ≥2.0 liter-per-minute pm home oxygen requirement
* An estimated Left Ventricular Ejection Fraction ≤40% (echo or MUGA)
* Hepatic cirrhosis (Biopsy Proven)
* HIV positive, ineligible because of the increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Pregnant or breastfeeding women are excluded from this study because the immunomodulatory treatment, preparative regimen, and anti-GVHD therapy contain agents with the potential for teratogenic or abortifacient effects.
* Evidence of uncontrolled bacterial, viral, or fungal infections (currently taking medication and progression of clinical symptoms) within 1 month prior to starting the conditioning regimen. Patients with fever or suspected minor infection should await resolution of symptoms before starting the conditioning regimen.
* Prior allogeneic marrow or stem cell transplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Probability of Engraftment | 42 Days after transplant
  The number of patients with engraftment (as defined as recovery of ANC to 500 cells per cubic mm) compared to the total number of patients treated as a function of the patient's age.

SECONDARY OUTCOMES:
Mean time to engraftment | 42 Days after transplant
  The average time to for engraftment (as defined as recovery of ANC to 500 cells per cubic mm) to occur estimated using a Kaplan-Meier curve as a function of the patient's age.
Disease Progression | 1 year
  The average time (in days) to disease progression estimated using a Kaplan-Meier curve
Overall Survival | 1 year
  The average time (in days) patients are alive after treatment estimated using a Kaplan-Meier curve
Follicular Stimulating Hormone Levels | 1 year
  Estimated difference in changes in Follicular Stimulating Hormone Levels after transplant, among patients with matched sibling donors compared to patients with alternate donors.
Luteinizing Hormone Levels | 1 year
  Estimated difference in changes in Luteinizing hormone Levels after transplant, among patients with matched sibling donors compared to patients with alternate donors.
Testosterone Levels | 1 year
  Estimated difference in changes in Testosterone Levels after transplant, among male patients with matched sibling donors compared to patients with alternate donors.
Graft versus Host Disease | 1 year
  The number patients with Grade III-IVGraft versus Host Disease as defined by CTCAE v4.0 in matched sibling compared to alternate-donor graft recipients
Cerebral Vasculopathy | 1 year
  Vasculopathy may clinically manifest as a history of stroke. The difference in number of strokes before and after transplantation will be evaluated with paired statistical tests (t-test or McNemar).
Renal Vasculopathy | 1 year
  Vasculopathy may clinically manifest as macroalbuminuria (≥300mg/g urinary albumin-to-creatinine ratio) or as a depressed estimated glomerular flow rate (eGFR). Evidence of renal vasculopathy before and after transplantation will be evaluated with paired statistical tests (t-test or McNemar).
Pulmonary Vasculopathy | 1 year
  Vasculopathy may clinically manifest as pulmonary arterial systolic pressure (PASP) by echo. Difference in PASP levels before and after transplantation will be evaluated with paired statistical tests (t-test or McNemar).
Hematopoiesis | 1 year
  Levels of stress hematopoiesis will be assessed by measuring telomere lengths with PCR before and after transplantation. These levels will be evaluated with paired statistical tests (t-test or McNemar).
Erythropoiesis | 1 year
  Levels of stress erythropoiesis will be assessed by measuring telomere lengths with PCR before and after transplantation. These levels will be evaluated with paired statistical tests (t-test or McNemar).

CONTACTS AND LOCATIONS:
Overall Officials: Molly Gallogly, MD, PhD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States